CLINICAL TRIAL: NCT06990971
Title: Harnessing the Disease Signatures From Endometrium and Menstrual Blood to Identify Avenues for the Treatment of Chronic Conditions Such as Endometriosis and Related Pathologies
Brief Title: Harnessing the Disease Signatures From Endometrium and Menstrual Blood to Identify Avenues for the Treatment of Chronic Conditions Such as Endometriosis and Related Pathologies: This is an Observational Study Aimed at Shedding Light on Women's Health
Acronym: CYCLE_ENDO
Status: Not yet recruiting | Type: Observational
Sponsor: Cycle Therapeutics Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: CYCLETX_OBS_REC_001
Record Dates: First submitted 2025-05-18; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Endometriosis; Infertility; Endometrial Cancer; Adenomyosis, Endometriosis
Keywords: Menstrual Fluid; Endometriosis; Tissue modelling
MeSH Terms: conditions — Endometriosis; Infertility; Endometrial Neoplasms; Adenomyosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Biospecimen Retention: Samples With DNA — Menstrual Tissue and biopsies will be stored frozen or fixed whole. This includes whole blood, tissue chunks and cells. DNA, RNA and protein may be extracted from the stored samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Endometriosis patients: Participants that have had a definitive diagnosis for endometriosis, often through laparoscopic surgery
  Interventions: Other: No Intervention: Observational Cohort
- Control: Participants that do not experience any gynaecological symptoms and have not been diagnoses with any gynaecological condition.
  Interventions: Other: No Intervention: Observational Cohort
- Symptomatic: Participants that may not have an endometriosis diagnosis, but have another diagnosed condition or display symptoms of endometriosis or dysmenorrhea.
  Interventions: Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: No Intervention: Observational Cohort — No interventions will be performed specifically for this study. Samples will be collected from menstrual fluid naturally shed or from biopsies and/or operations that are already taking place.

SUMMARY:
Many women's health conditions have limited treatments available and poor outcomes, in part due to the lack of understanding of disease processes and lack of data available. This study aims to build knowledge in women's health by leveraging the information we can gather from menstrual fluid and the uterus. By looking at samples from menstrual fluid and biopsies and associating it with health outcomes of the people donating these samples, we will be able to find new signatures of disease. This can help us find early diagnostic markers, better classify diseases and give us the tools that allow us to build the right models in the lab to find new treatments. By collecting this data, we will be able to identify patterns within given diseases that can help us cure them and derive the cells necessary to model the disease. The study is funded and undertaken by Cycle Therapeutics, a company with the mission of curing endometriosis. All women above the age of 16 will be eligible, although most samples will be collected from those who are menstruating or already undergoing biopsies/surgical tissue removal. Women with endometriosis or suspicion of the disease are encouraged to take part, but participation of people without any symptoms or conditions is important to understand what the base healthy state looks like. Most of the sample processing will be done within Cycle and collection will occur at clinics or remotely, and can be as simple as pouring menstrual fluid from a cup into a tube to ship to Cycle. The study will last four years, during which we hope to build a strong understanding of conditions affecting women. We will be able to provide health insight to donors after each donation, but the greatest value in this study will lie in the new treatments we can discover thanks to our novel understanding.

ELIGIBILITY:
Inclusion Criteria:

* Menstruating

Exclusion Criteria:

* Not menstruating

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All women above the age of 16 will be eligible, although most samples will be collected from those who are menstruating. Women with endometriosis or suspicion of the disease are encouraged to take part, but participation of people without any symptoms or conditions is important to understand what the base healthy state looks like. Because we are trying to broadly understand women's health, we welcome participation of females across all conditions.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2029-05-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Identifying tissue signatures of endometriosis | 1-4 years
  The principal research objective is to identify signatures of endometriosis within the samples collected. These signatures can help us understand:
  1. - Whether endometriosis is one disease or many sub-diseases, therefore informing how we treat each patient.
  2. - What endometriosis tissue looks like. This will be used to build our lab models that we will use to test therapies on.
  3. - What drives progression of the disease. Recurrent measurements will allow us to tease out which processes are involved in disease progression.
  4. - How endometriosis cells compare to control cells in a dish. This will be critical to establishing the right read outs for our search of novel drugs that can reverse the disease.

SECONDARY OUTCOMES:
The value of menstrual fluid in health research | 1-4 years
  When collecting the clinical and biological data from donors, we may be able to identify early diagnostic markers of certain particular conditions, or predict the prognosis of others. We may also find a very robust signature of another disease related or unrelated to endometriosis. Our aim is to more broadly assess the descriptive value of menstrual fluid and tissue biopsies.
Menstrual cell potential | 1-4 years
  We will determine the value of cells isolated from menstrual fluid and biopsies in both disease modelling and therapeutic interventions.

IPD SHARING:
Plan to Share IPD: No
Given the collection of menstrual fluid will occur outside of a primary care centre, personal data will have to be anonymised directly by the company receiving these samples. This will be made clear to participants in the consent form.
  Personally identifiable information will only be accessible by a restricted and trained group of people within the organisation or working closely with it.
  Analysts from Cycle Therapeutics will only analyse pseudonymised data. Where third parties are employed in the recruitment of participants, they will only be able to access pseudonymised information.
  Where appropriate, anonymised data will be shared with collaborators and partners of Cycle Therapeutics, ensuring that there is no way to identify the participants through this information.

REFERENCES:
- See also: The web page for more information and to sign up to donate menstrual fluid — https://www.cycletherapeutics.org/donate-menstrual-fluid